CLINICAL TRIAL: NCT01512992
Title: Renewing Health RCT in Catalonia for the Evaluation of Home Telehealth Follow-up After Hospital Discharge for COPD Patients
Brief Title: Home Telehealth Follow-up After Hospital Discharge for Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catalan Agency for Health Information, Assessment and Quality (Other Government)
Collaborators: Fundació TicSalut (Other); Hospital Clinic of Barcelona (Other); Hospital de Mataró (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RH_pilotCAT; EC Grant Agreement 250487 (Other Grant/Funding Number: European Comission, Information Society and Media DG)
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home telehealth (Experimental)
  Interventions: Procedure: Home telehealth
- Usual care (No Intervention)

INTERVENTIONS:
Procedure: Home telehealth — Patients receive tailored intervention according to their clinical complexity.
  All patients in the intervention group receive:
  * Personalised care plan
  * Education on self-management
  * Access to a personalized online health folder
  * Access to Call center
  * Access to primary care and hospital specialists; follow-up visits for evaluation of clinical recovery and care plan adjustments (if needed).
  Patients with LOW complexity additionally receive:
  * Daily videoconferences for the 1st week after discharge
  * Remote monitoring for respiratory parameters. Sensors are selected on an individual basis by the medical specialists.
  Patients with HIGH complexity additionally receive:
  * Videoconferences for at least 1 month after discharge, scheduled on an individual basis.
  * Remote monitoring for respiratory parameters.
  * One monthly phone call from the call centre to promote and assess patient self-management.
  Arms: Home telehealth

SUMMARY:
The purpose of this study is to assess the effects of a complex telemedicine intervention as a part of an integrated care program for patients with chronic obstructive pulmonary disease (COPD) discharged from the hospital after disease exacerbation. Will be evaluated whether the intervention produces benefits in terms of mortality, reduction in hospital readmissions and health-related quality of life. In addition, the trial evaluates the economical and organizational impact of the new service and examines its acceptability by patients and health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Exacerbation of COPD
* Age > 40 years
* Capability to use the devices provided
* Willing to participate

Exclusion Criteria:

• Participation in a previous COPD home telehealth study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of hospital readmissions | 3 months period

SECONDARY OUTCOMES:
Health related quality of life of the patients as measured by the SF-36 v2 questionnaire | 3 months - at baseline and study end
Hospital anxiety and depression scale HADS | 3 months - at baseline and study end
Lung condition as measured by FEV1 | 3 months - at baseline and study end
Condition-related health status measured by COPD Assessment Test (CAT) | 3 months - at baseline and study end
Mortality | 3 months period
Patients' Acceptance-Satisfaction measured by the WSD Questionnaire | at the 3rd month of the telehealth intervention
Time in days to first readmission | 3 months period
Length of stay in days for each readmission | 3 months period
Number of emergency room visits | at the 3rd month (end of trial)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Roca Torrent, MD, Principal Investigator — Pulmonary Department - Hospital Clinic of Barcelona
Locations (8):
- Spain (8):
  - Hospital Germans Trias i Pujol, Badalona, Catalonia
  - Capio Hospital Universitari Sagrat Cor, Barcelona, Catalonia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Plató, Barcelona, Catalonia
  - Hospital de Mataró, Mataró, Catalonia
  - Hospital Parc Taulí, Sabadell, Catalonia
  - Consorci Sanitari de Terrassa, Terrassa, Catalonia

REFERENCES:
- [Background] Casas A, Troosters T, Garcia-Aymerich J, Roca J, Hernandez C, Alonso A, del Pozo F, de Toledo P, Anto JM, Rodriguez-Roisin R, Decramer M; members of the CHRONIC Project. Integrated care prevents hospitalisations for exacerbations in COPD patients. Eur Respir J. 2006 Jul;28(1):123-30. doi: 10.1183/09031936.06.00063205. Epub 2006 Apr 12. PMID 16611656
- [Background] Finkelstein SM, Speedie SM, Potthoff S. Home telehealth improves clinical outcomes at lower cost for home healthcare. Telemed J E Health. 2006 Apr;12(2):128-36. doi: 10.1089/tmj.2006.12.128. PMID 16620167
- [Background] Polisena J, Tran K, Cimon K, Hutton B, McGill S, Palmer K, Scott RE. Home telehealth for chronic obstructive pulmonary disease: a systematic review and meta-analysis. J Telemed Telecare. 2010;16(3):120-7. doi: 10.1258/jtt.2009.090812. Epub 2010 Mar 2. PMID 20197355